CLINICAL TRIAL: NCT05098249
Title: Ferric Carboxymaltose With or Without Phosphate Substitution for the Treatment of Iron Deficiency or Iron Deficiency Anemia Before Elective Surgery - the DeFICIT Trial
Brief Title: Ferric Carboxymaltose With or Without Phosphate Substitution for the Treatment of Iron Deficiency or Iron Deficiency Anemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Donat R. Spahn (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor-Investigator, Donat R. Spahn, Prof. Dr. med., University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-00383
Record Dates: First submitted 2021-10-14; First posted 2021-10-28 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Anemia; Iron-deficiency; Hypophosphatemia
Keywords: iron-deficiency anemia; hypophosphatemia; elective surgery; iron-deficiency; preoperative iron substitution; phosphate substitution
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency; Hypophosphatemia | interventions — calcium D-pantothenate, L-cysteine drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum (Experimental)
  Interventions: Drug: Verum
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Verum — The participant takes two capsules Phoscap® (3mmol/capsule) orally three times a day over 30 days beginning the day of Ferinject administration.
  Arms: Verum
Drug: Placebo — The participant takes wo capsules Placebo orally three times a day over 30 days beginning the day of Ferinject administration.
  Arms: Placebo

SUMMARY:
This is a confirmatory trial to establish superior serum phosphate stability associated with use of Phoscap® compared with placebo as a supplement for treatment of iron deficiency or iron deficiency anemia with Ferinject® before elective surgery.

DETAILED DESCRIPTION:
Iron deficiency anemia is a global health problem most commonly caused by excessive blood loss, impaired intestinal iron absorption, or chronic inflammation. In the perioperative setting, intravenous ferric carboxymaltose allows efficient treatment of preoperative iron deficiency and anemia. Recent studies have implied that ferric carboxymaltose might cause hypophosphatemia. Notably, hypophosphatemia has been associated with less muscle strength, which may influence early post-surgery recovery of patients. Additional oral phosphate supplementation may alleviate this hypophosphatemia.

This is a confirmatory trial to establish superior serum phosphate stability associated with use of Phoscap® compared with placebo as a supplement for treatment of iron deficiency or iron deficiency anemia with Ferinject® before elective surgery.

This is also a confirmatory trial to establish non-inferior efficacy of Phoscap® compared with placebo for the treatment of iron deficiency or iron deficiency anemia with Ferinject®; and to establish superior core muscle strength associated with the use of Phoscap® compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix 5: Informed Consent Form)
* Male or female ASA 1 to 3 patients, at least 18 years old
* Scheduled for an elective major abdominal or thoracic surgery.
* Patients with isolated iron deficiency (defined as hemoglobin concentration (Hb) > 130 g/l, and plasma Ferritin < 100 ng/ml or TSAT < 20%), or iron deficiency anemia (defined as Hb 100-130 g/l, and plasma Ferritin < 100 ng/ml or TSAT < 20%).
* Patients scheduled to be hospitalized ≥ 3 days.

Exclusion Criteria:

* Patients with known anaphylactic reactions to parenteral iron products. Patients with allergy/hypersensitivity to any contents of Ferinject® or Phoscap®.
* Patients with iron overload or disturbances in utilization of iron (e.g. haemochromatosis, hemosiderosis).
* Patients with ≥3 times increase in aspartate aminotransferase or alanine aminotransferase as per reference range.
* Patients with excessive blood loss requiring massive transfusion (≥ 10 more red blood cell units).
* Patients with known myelodysplastic syndromes.
* Patients with chronic kidney disease with an estimated GFR < 30 ml/min or with end-stage renal disease requiring scheduled dialysis.
* Patients with known urinary tract infections with urea-splitting bacteria.
* Patients with known diseases influencing phosphate, calcium or vitamin D homeostasis (e.g. Hyperparathyroidism, X-linked hypophosphatemia, renal tubular acidosis).
* Patients taking medication significantly influencing phosphate, calcium or vitamin D homeostasis (e.g. vitamin D substitution > 800 I.E. per day in the last 4 months, pre-existing phosphate substitution, phosphate binders).
* Patients with preexisting hypophosphatemia
* Any patient judged to lack the ability to give informed consent or perform the trial assessments (e.g. due to dementia, insufficient knowledge of the German language).
* Women who are pregnant or breast feeding,
* Intention to become pregnant during the course of the study,
* Lack of safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases (Female participants who are surgically sterilized / hysterectomized or post-menopausal for longer than 2 years are not considered as being of child bearing potential),
* Known or suspected non-compliance, drug or alcohol abuse.
* Participation in another study with investigational drug within the 30 days preceding and during the present study.
* Any patient judged by the Principal Investigator or Sub-Investigator to be inappropriate for the trial for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Establish superior serum phosphate stability | 3 years
  The primary endpoint is superior serum phosphate stability. The investigators measure perioperative phosphate concentrations in participants during the follow-up visits and compare the results between verum and placebo group.

SECONDARY OUTCOMES:
Perioperative hemoglobin concentration | 3 years
  Mean perioperative Hb of the day of surgery, post-operative day (POD)2 and POD4.
Core muscle strength | 3 years
  Pre- and postoperative assessment of core muscle strength by volitional testing of maximal inspiratory and expiratory pressures.

CONTACTS AND LOCATIONS:
Overall Officials: Donat R Spahn, Prof. Dr., Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Munoz M, Gomez-Ramirez S, Campos A, Ruiz J, Liumbruno GM. Pre-operative anaemia: prevalence, consequences and approaches to management. Blood Transfus. 2015 Jul;13(3):370-9. doi: 10.2450/2015.0014-15. Epub 2015 Jun 16. No abstract available. PMID 26192787
- [Result] Munoz M, Laso-Morales MJ, Gomez-Ramirez S, Cadellas M, Nunez-Matas MJ, Garcia-Erce JA. Pre-operative haemoglobin levels and iron status in a large multicentre cohort of patients undergoing major elective surgery. Anaesthesia. 2017 Jul;72(7):826-834. doi: 10.1111/anae.13840. Epub 2017 Apr 6. PMID 28382661
- [Result] Wolf M, Koch TA, Bregman DB. Effects of iron deficiency anemia and its treatment on fibroblast growth factor 23 and phosphate homeostasis in women. J Bone Miner Res. 2013 Aug;28(8):1793-803. doi: 10.1002/jbmr.1923. PMID 23505057